CLINICAL TRIAL: NCT01387230
Title: A12-Week, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of GSK573719 Delivered Once-Daily Via a Novel Dry Powder Inhaler in Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: Evaluate the Efficacy and Safety of GSK573719 Delivered Via a Novel Dry Powder Inhaler in Subjects With COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 115408
Record Dates: First submitted 2011-06-30; First posted 2011-07-04 (Estimated); Results first posted 2014-02-11 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: chronic obstructive pulmonary disease; long acting muscarinic antagonist
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — GSK573719

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK573719 (Experimental): active drug
  Interventions: Drug: GSK573719
- Placebo (Placebo Comparator): no active drug
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GSK573719 — 62.5 mcg
  Arms: GSK573719
Drug: GSK573719 — 125mcg
  Arms: GSK573719
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess if 12 weeks' treatment with GSK573719 Inhalation Powder is safe and effective compared with placebo or no active drug intake, when administered once-daily in subjects with Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
Inhaled bronchodilators, such as beta 2 agonists and anticholinergics, and inhaled corticosteroids are the mainstays of therapy in patients diagnosed with COPD. Anticholinergic bronchodilators or long acting muscarinic receptor antagonists function by blocking endogenous airway smooth muscle cholinergic tone. Treatment with anticholinergics has been shown to significantly improve forced expiratory volume in 1 second (FEV1), resting and dynamic lung hyperinflation, symptoms, and exercise capacity in patients with COPD. Currently tiotropium is the only approved long acting muscarinic antagonist available for treatment of COPD.This is a multicenter, randomized, double-blind, placebo-controlled, parallel group study to evaluate the efficacy and safety of GSK573719 Inhalation Powder of 2 doses when administered once-daily via Novel DPI compared with placebo over a treatment period of 12 weeks in subjects with COPD. There will be a total of 8 study clinic visits conducted on an outpatient basis. Subjects who meet the eligibility criteria at Screening (Visit 1) will complete a 5 to 9 days run-in period followed by a 12-week treatment period. There will be 8 clinic visits during three of which serial spirometry will be performed . The total duration of subject participation in the study will be approximately 14 weeks.

This is a Phase III multicenter, randomized, double-blind, placebo-controlled, parallel group study to evaluate the efficacy and safety of GSK573719 Inhalation Powder 62.5 mcg and 125 mcg when administered once-daily via Novel DPI compared with placebo over a treatment period of 12 weeks in subjects with COPD.

Eligible subjects will be randomized 1:1:1 to receive either of the two doses of GSK573719 Inhalation Powder doses or placebo for 12 weeks.

There will be a total of 8 study clinic visits conducted on an outpatient basis. Subjects who meet the eligibility criteria at Screening (Visit 1) will complete a 5 to 9 days run-in period followed by a 12-week treatment period. Clinic visits will be at Screening, Randomization (Visit 2), Day 3 and Weeks 2, 4, 8, and 12, and 1 day after the Week 12 visit (Visits 1 to 8, respectively). A safety follow-up assessment will be conducted by telephone approximately 7 days after the end of the study treatment (FU Phone Contact). The total duration of subject participation, including the follow-up period will be approximately 14 weeks. All subjects will be provided with albuterol/salbutamol for use on an "as-needed" basis throughout the run-in and treatment periods.

Pre-dose spirometry will be conducted at each clinic visit. Six hour post-dose serial spirometry will be conducted at Visit 2 and at Visits 5 and 7. All subjects will be provided with a paper diary for completion everyday throughout the run-in period and 12-week treatment period. Subjects will use the diary to record their daily use of supplemental albuterol/salbutamol and to record any medical problems experienced and any medications used.

At Visit 2 the Baseline Dyspnea Index (BDI) will be administered. The Transition Dyspnea Index (TDI) will be administered at Visits 5, 6, and 7.

Disease specific health status will be evaluated using the St. George's Respiratory Questionnaire (SGRQ) at Visit 2 and Visits 5, 6 and 7. Vital signs (blood pressure and pulse rate), 12-lead ECGs and standard clinical laboratory tests (hematology and blood biochemistry) including pharmacokinetic samples will be obtained at selected clinic visits.

Approximately 198 subjects will be randomized to ensure at least 168 subjects complete the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD
* 10 pack-year or greater history of cigarette smoking
* Post-bronchodilator FEV1/FVC of <0.7
* Predicted FEV1 of 70% of normal or less
* Modified Medical Research Council (mMRC) dyspnea score of 2 or greater

Exclusion Criteria:

* Women who are pregnant, lactating, or planning to become pregnant
* Respiratory disorders other than COPD, including a current diagnosis of asthma
* Clinically significant non-respiratory diseases or abnormalities that are not adequately controlled
* Significant allergy or hypersensitivity to anticholinergics, beta2-agonists, or the excipients of magnesium stereate or lactose used in the inhaler delivery device
* Hospitalization for COPD or pneumonia within 12 weeks prior to screening
* Lung volume reduction surgery within 12 weeks prior to screening
* Abnormal and clinically significant ECG findings at screening
* Clinically significant laboratory findings at screening
* Use of systemic corticosteroids, antibiotics for respiratory tract infections, high dose inhaled steroids (>1000mcg fluticasone propionate or equivalent), PDE4 inhibitors, tiotropium, oral beta2-agoinists, short- and long-acting inhaled beta2-agonists, inhaled sodium cromoglycate or nedocromil sodium, or investigational medicines for defined time periods prior to the screening visit
* Use of long-term oxygen therapy (12 hours or greater per day)
* Regular use of nebulized treatment with short-acting bronchodilators
* Participation in the acute phase of a pulmonary rehabilitation program
* A know or suspected history of alcohol or drug abuse
* Affiliation with the investigational site
* Previous use of GSK573719 or the combination of GSK573719/GW642444

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2011-07-01; Primary Completion 2012-02-01 (Actual); Study Completion 2012-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (23):
- United States (4):
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Easley, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina
- Germany (14):
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Gelnhausen, Hesse
  - GSK Investigational Site, Kassel, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Weyhe-Leeste, Lower Saxony
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Solingen, North Rhine-Westphalia
  - GSK Investigational Site, Koblenz, Rhineland-Palatinate
  - GSK Investigational Site, Leipzg, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Teuchern, Saxony-Anhalt
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Berlin
- Japan (5):
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Trivedi R, Richard N, Mehta R, Church A. Umeclidinium in patients with COPD: a randomised, placebo-controlled study. Eur Respir J. 2014 Jan;43(1):72-81. doi: 10.1183/09031936.00033213. Epub 2013 Aug 15. PMID 23949963
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 115408 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115408 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115408 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115408 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115408 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115408 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115408 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (par.) who met eligibility criteria at Screening (Visit 1) completed a 5- to 9-day run-in period and were then randomized to a 12-week treatment period. A total of 246 par. were screened; 206 par. who were eligible were randomized and 206 par. received at least one dose of study drug.
Groups:
- Placebo: Participants received matching placebo once daily (QD) via a dry powder inhaler (DPI) in the morning for 12 weeks.
- UMEC 62.5 µg QD: Participants received umeclidinium bromide (UMEC) 62.5 micrograms (µg) QD via a DPI in the morning for 12 weeks.
- UMEC 125 µg QD: Participants received UMEC 125 µg QD via a DPI in the morning for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | UMEC 62.5 µg QD | UMEC 125 µg QD
Started | 68 | 69 | 69
Completed | 50 | 62 | 56
Not Completed | 18 | 7 | 13
Not completed — Adverse Event | 0 | 1 | 3
Not completed — Lack of Efficacy | 8 | 5 | 4
Not completed — Protocol-defined Stopping Criteria | 6 | 0 | 5
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants received matching placebo QD via a DPI in the morning for 12 weeks.
- UMEC 62.5 µg: Participants received UMEC 62.5 µg QD via a DPI in the morning for 12 weeks.
- UMEC 125 µg: Participants received UMEC 125 µg QD via a DPI in the morning for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | UMEC 62.5 µg | UMEC 125 µg | Total
Number analyzed (Participants) | 68 | 69 | 69 | 206
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.5 (8.72) | 62.3 (9.50) | 64.6 (7.96) | 63.1 (8.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 27 | 78
  Male | 42 | 44 | 42 | 128
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 1 | 1 | 2 | 4
  Asian - Japanese Heritage | 8 | 7 | 6 | 21
  White - Arabic/North African Heritage | 1 | 1 | 0 | 2
  White - White/Caucasian/European Heritage | 58 | 60 | 61 | 179

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (BL) in Trough Forced Expiratory Volume in One Second (FEV1) on Day 85
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 measurements were taken electronically by spirometry on Days 2, 14, 28, 56, 84, and 85. Baseline is defined as the mean of the assessments made 30 minutes pre-dose and 5 minutes pre-dose on Treatment Day 1. Trough FEV1 is defined as the mean of the FEV1 values obtained at 23 and 24 hours after the previous morning's dosing (ie., trough FEV1 on Day 85 is the mean of the FEV1 values obtained 23 and 24 hours after the morning dosing on Day 84). Change from Baseline was calculated as the trough FEV1 minus the Baseline. Analysis was performed using a repeated measures model with covariates of treatment, Baseline , smoking status, center group, day, and day by Baseline and day by treatment interactions.
Time Frame: Baseline and Day 85
Population: Intent-to-Treat (ITT) Population: all randomized par. who received >=1 dose of study drug. Par. analyzed are those with data available at the presented time point; but, all par. without missing covariate information and with >=1 post-BL measurement were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | UMEC 62.5 µg | UMEC 125 µg
Number analyzed (Participants) | 50 | 61 | 55
Liters | -0.007 (0.0280) | 0.120 (0.0257) | 0.145 (0.0268)
Statistical Analysis 1: Comparison: Placebo vs UMEC 62.5 µg; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.127, 95% CI 2-sided [0.052 to 0.202] — Least squares mean difference=UMEC 62.5 µg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs UMEC 125 µg; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Restricted maximum likelihood (REML)-based repeated measures approach (MMRM); Least squares mean difference = 0.152, 95% CI 2-sided [0.076 to 0.229] — Least squares mean difference=UMEC 125 µg minus Placebo

2. Secondary Outcome: Change From Baseline in Weighted Mean (WM) 0-6 Hour FEV1 Obtained Post-dose at Days 1, 28 (Week 4) and 84 (Week 12)
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. The WM FEV1 was derived by calculating the area under the FEV1/time curve (AUC) using the trapezoidal rule, and then dividing the value by the time interval over which the AUC was calculated. The WM was calculated at Days 1, 28, and Day 84 using the 0-6-hour post-dose FEV1 measurements collected on that day, which included pre-dose (Day 1: 30 minutes [min] and 5 min prior to dosing; other serial visits: 23 and 24 hours after the previous morning dose) and post-dose at 1 hour, 3 hours, and 6 hours. Change from Baseline was the WM minus Baseline. Analysis was performed using a repeated measures model with covariates of treatment, Baseline (mean of the two assessments made 30 minutes and 5 minutes pre-dose on Day 1), smoking status, center group, day, and day by Baseline and day by treatment interactions.
Time Frame: Baseline and Days 1, 28 and 84
Population: ITT Population. All participants with >=1 post-BL assessment and non-missing covariate data are included in the analysis. Different participants may have been analyzed at different time points (represented by n=X, X, X in the category titles), so the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | UMEC 62.5 µg | UMEC 125 µg
Number analyzed (Participants) | 68 | 69 | 69
Liters
  Day 1, n=66, 69, 69 | 0.017 (0.0150) | 0.141 (0.0147) | 0.164 (0.0147)
  Day 28, n= 53, 65, 60 | -0.024 (0.0223) | 0.141 (0.0206) | 0.172 (0.0212)
  Day 84, n= 49, 60, 56 | -0.003 (0.0271) | 0.163 (0.0248) | 0.188 (0.0256)

3. Secondary Outcome: Change From Baseline in Serial FEV1 Over 24 Hours Post-dose at Days 1 and 84 (Week 12)
Description: Pulmonary function was measured by FEV1, defined as the maximal amount of air that can be forcefully exhaled in one second. Serial FEV1 measurements were taken electronically by spirometry. Serial FEV1 measurements of interest for Day 1 were collected at 1, 3, 6, 23 and 24 hours post-dose on Day 1 and for Day 84, the measures were pre-dose (24 hours post-dose of Day 83 morning dose but prior to Day 84's dose) and 1, 3, 6, 23 and 24 hours post dose on Day 84. Baseline is the mean of the two assessments made 30 minutes and 5 minutes pre-dose on Day 1. Change from Baseline was calculated as FEV1 value at the evaluated time point minus Baseline. Analysis performed separately by Visit/Day using a repeated measures model with covariates of treatment, Baseline, smoking status, center group, time, time by Baseline and time by treatment interactions.
Time Frame: Baseline, Day 1 and Day 84
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | UMEC 62.5 µg | UMEC 125 µg
Number analyzed (Participants) | 68 | 69 | 69
Liters
  Day 1, 1 hour, n=68, 69, 69 | -0.001 (0.0148) | 0.132 (0.0147) | 0.142 (0.0147)
  Day 1, 3 hours ,n=68, 69, 69 | 0.035 (0.0187) | 0.165 (0.0186) | 0.210 (0.0186)
  Day 1, 6 hours, n=66, 69, 69 | 0.000 (0.0206) | 0.156 (0.0203) | 0.169 (0.0203)
  Day 1, 23 hours, n=67, 69, 65 | -0.027 (0.0178) | 0.070 (0.0176) | 0.113 (0.0180)
  Day 1, 24 hours, n=67, 69, 66 | -0.020 (0.0190) | 0.099 (0.0188) | 0.151 (0.0191)
  Day 84, Pre-dose, n=50, 60, 56 | 0.002 (0.0299) | 0.155 (0.0269) | 0.177 (0.0283)
  Day 84, 1 hour,n=50, 60, 56 | -0.025 (0.0299) | 0.167 (0.0270) | 0.199 (0.0283)
  Day 84, 3 hours, n=50, 61, 56 | 0.012 (0.0301) | 0.189 (0.0271) | 0.219 (0.0285)
  Day 84, 6 hours,n=49, 61, 56 | 0.006 (0.0286) | 0.159 (0.0257) | 0.178 (0.0270)
  Day 84, 23 hours, n=50, 60, 55 | -0.019 (0.0301) | 0.106 (0.0271) | 0.142 (0.0286)
  Day 84, 24 hours, n=50, 61, 55 | 0.020 (0.0299) | 0.142 (0.0269) | 0.170 (0.0284)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study medication until the end of treatment (up to 12 weeks).
Description: SAEs and non-serious AEs were collected in members of the ITT Population, comprised of all participants who had received at least one dose of randomized study medication during treatment period.
Arm/Group | Placebo | UMEC 62.5 µg | UMEC 125 µg
Serious Adverse Events (participants affected / at risk) | 1/68 | 1/69 | 2/69
Other Adverse Events (participants affected / at risk) | 16/68 | 12/69 | 19/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=68) | UMEC 62.5 µg (N=69) | UMEC 125 µg (N=69)
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=68) | UMEC 62.5 µg (N=69) | UMEC 125 µg (N=69)
Nasopharyngitis (Infections and infestations) | 7 | 8 | 7
Headache (Nervous system disorders) | 7 | 5 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.